CLINICAL TRIAL: NCT02458417
Title: Autologous Cell Suspension Grafting Using ReCell in Vitiligo and Piebaldism Patients: a Randomized Controlled Study on the Recipient Site Preparation
Brief Title: Autologous Cell Suspension Grafting Using ReCell in Vitiligo and Piebaldism Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Netherlands Institute for Pigment Disorders (Other)
Collaborators: Avita Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL49720.018.14
Record Dates: First submitted 2015-05-26; First posted 2015-06-01 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2015-05

CONDITIONS: Segmental Vitiligo; Piebaldism
Keywords: Ablative laser; Fractional laser; Vitiligo; Piebaldism; Cell suspension grafting
MeSH Terms: conditions — Piebaldism; Vitiligo

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Full surface CO2 laser 200mJ + ReCell (Active Comparator): This test region will receive full surface pretreatment with the CO2 laser (Ultrapulse, ActiveFX handpiece, Lumenis Inc., Santa Clara, CA, USA) at 200 mJ (depth 209 µm) and density 3. After pretreatment ReCell autologous epidermal cell suspension will be applied on this test region.
  Interventions: Device: ReCell; Device: Full surface CO2 laser 200 mJ
- Full surface CO2 laser 150mJ + ReCell (Experimental): This test region will receive full surface pretreatment with the CO2 laser (Ultrapulse, ActiveFX handpiece, Lumenis Inc., Santa Clara, CA, USA) at 150 mJ (depth 144 µm) and density 3. After pretreatment ReCell autologous epidermal cell suspension will be applied on this test region.
  Interventions: Device: ReCell; Device: Full surface CO2 laser 150 mJ
- Fractional CO2 laser 7.5mJ 20% + ReCell (Experimental): This test region will receive pretreatment with the fractional CO2 laser (Ultrapulse, DeepFX handpiece, Lumenis Inc., Santa Clara, CA, USA) at 7.5 mJ/microbeam (depth 225 µm) and 20% density. After pretreatment ReCell autologous epidermal cell suspension will be applied on this test region.
  Interventions: Device: ReCell; Device: Fractional CO2 laser 7.5 mJ, 20%
- Control (No Intervention): No intervention

INTERVENTIONS:
Device: ReCell — A split-thickness skin biopsy will be taken from the hip region of the patient. The skin biopsy that is obtained will be treated in the ReCell kit (Avita Medical Europe Ltd, Cambridge, UK): it will be placed in the heated enzyme solution, containing trypsin, in the device for 15-20 minutes to allow cell disaggregation. After that period, the biopsy will be taken from the enzyme solution and will be dipped in sodium lactate buffer solution. The biopsy will then be scraped to disaggregate the cells from the dermal epidermal junction. The epidermal cells are drawn up in a syringe. The prepared suspension will be dripped on both donor and acceptor site.
  Other Names: ReCell autologous cell suspension grafting
  Arms: Fractional CO2 laser 7.5mJ 20% + ReCell; Full surface CO2 laser 150mJ + ReCell; Full surface CO2 laser 200mJ + ReCell
Device: Full surface CO2 laser 200 mJ — Full surface pretreatment with the CO2 laser (Ultrapulse, ActiveFX handpiece, Lumenis Inc., Santa Clara, CA, USA) at 200 mJ (depth 144 µm) and density 3
  Arms: Full surface CO2 laser 200mJ + ReCell
Device: Full surface CO2 laser 150 mJ — Full surface pretreatment with the CO2 laser (Ultrapulse, ActiveFX handpiece, Lumenis Inc., Santa Clara, CA, USA) at 150 mJ (depth 144 µm) and density 3
  Arms: Full surface CO2 laser 150mJ + ReCell
Device: Fractional CO2 laser 7.5 mJ, 20% — Pretreatment with the fractional CO2 laser (Ultrapulse, DeepFX handpiece, Lumenis Inc., Santa Clara, CA, USA) at 7.5 mJ/microbeam (depth 225 µm) and 20% density.
  Arms: Fractional CO2 laser 7.5mJ 20% + ReCell

SUMMARY:
The purpose of this study is to assess the efficacy and safety of ReCell grafting after CO2 laser abrasion with superficial full surface ablation, fractional laser treatment and conventional (deep) full surface CO2 laser ablation, to assess the practical aspects and the patient reported outcome and to assess the cellular composition of the graft.

DETAILED DESCRIPTION:
Autologous epidermal cell suspension grafting is an effective method of surgical treatment in vitiligo, which is suitable for treating large areas with good cosmetic results. The ReCell Autologous Cell Harvesting Device (Avita Medical Europe Limited, Cambridge, UK) is a device which, compared to other forms of autologous epidermal cell suspension grafting, is easier in use showing similar results. With this device an epidermal cell suspension is created from a split skin graft, usually taken from the hip region. Currently, conventional ablative (full surface de-epidermisation) laser treatment in different laser settings is used as pre-treatment to prepare the acceptor site for transplantation. There is no evidence for the laser settings used and no studies are available on the use of a fractional laser as pre-treatment in autologous cell suspension grafting using ReCell (ReCell grafting). The investigators hypothesize that more superficial conventional ablative laser treatment and fractional ablative laser treatment are as effective as the current pre-treatment, whereas these treatments are less invasive, provide faster healing and prevent side effects like persisting erythema and scars. Furthermore, infiltration anaesthesia is not necessary with these less invasive treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patients with, segmental vitiligo or piebaldism under medical treatment at the Netherlands Institute for Pigment Disorders
* Age ≥18
* Patient is willing and able to give written informed consent
* Segmental vitiligo stable since 12 months without systemic therapy or 12 months without topical therapy as defined by the absence of new lesions and/or enlargement of existing lesions.
* At least four depigmented lesions on the proximal extremities or trunk larger than 3x3 cm or one depigmented lesion on the proximal extremities or trunk of at least 12x3 cm.

Exclusion Criteria:

* UV therapy or systemic immunosuppressive treatment during the last 12 months
* Local treatment of vitiligo during the last 12 months
* Vitiligo lesions with follicular or non-follicular repigmentations
* Skin type I
* Recurrent HSV skin infections
* Hypertrophic scars
* Keloid
* Cardiac insufficiency
* Patients with a history of hypersensitivity to (UVB or UVA) light and/or allergy to local anaesthesia.
* Patients who are pregnant or breast-feeding
* Patients not competent to understand what the procedures involves
* Patients with a personal history of melanoma or non-melanoma skin cancer
* Patients with atypical nevi.
* Known allergy to clarithromycin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-05; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Repigmentation | 6 months after intervention
  Assessment will be done by sheets and a digital image analysis system. To assess the pigmentation, the contours of pigmentation are copied on a transparent sheet before and six months after treatment, after which the sheets are scanned using a predefined resolution. By comparing pre- and post-treatment pictures, the relative surface showing repigmentation expressed as percentage of the selected treated patch are computed.

SECONDARY OUTCOMES:
PhGA | 6 months after intervention
  Blinded physician's assessment of repigmentation. Repigmentation will be classified as follows: 0-25%, 26-50%, 51-75%, 76-95%, 96-100% six months.
Side effects | 6 months after intervention
  Visual assessment of side effects per treatment region (erythema, hyperpigmentation, hypopigmentation and scar on a scale from 0-3) will be done by a blinded investigator six months.
Reepithelialization | 1 week after intervention
  One week after grafting reepithelialization will be assessed by a blinded physician and estimated on a 0 to 100% scale.
Colour difference | 6 months after intervention
  Colour difference i.e. the difference between normal pigmentation, erythema, and hyperpigmentation will be assessed with a DermaSpectrometer (Cortex Technology ApS, Hadsund, Denmark)
PGA | 6 months after intervention
  General outcome will be assessed by the patient per treatment region on a scale from 0-3 (Poor, Moderate, Good, and Excellent).
Pain | 1 week after intervention
  One week after grafting, pain will be assessed after grafting on a 100 mm visual analogue scale (VAS) per treatment region
Cell count | up to six hours
  The superfluous of the suspension will be used for flow cytometric analyses of the cellular composition of the graft.

OTHER OUTCOMES:
Skin type | week 0
  Fitzpatrick skin type
VIDA score | week 0
  Classification of disease activity according to VIDA scale
Duration of disease | week 0
  Duration of disease

CONTACTS AND LOCATIONS:
Overall Officials: Albert Wolkerstorfer, MD, PhD, Principal Investigator — Netherlands Institute for Pigment Disorders, Department of Dermatology, Academic Medical Center, University of Amsterdam; Menno A. De Rie, MD, PhD, Study Director — Department of Dermatology, Academic Medical Center, University of Amsterdam
Locations (1):
- Netherlands Institute for Pigment disorders, Amsterdam, Netherlands

REFERENCES:
- [Background] van Geel N, Ongenae K, Naeyaert JM. Surgical techniques for vitiligo: a review. Dermatology. 2001;202(2):162-6. doi: 10.1159/000051626. PMID 11306848
- [Background] Mulekar SV, Ghwish B, Al Issa A, Al Eisa A. Treatment of vitiligo lesions by ReCell vs. conventional melanocyte-keratinocyte transplantation: a pilot study. Br J Dermatol. 2008 Jan;158(1):45-9. doi: 10.1111/j.1365-2133.2007.08216.x. Epub 2007 Oct 10. PMID 17927795
- [Background] Manstein D, Herron GS, Sink RK, Tanner H, Anderson RR. Fractional photothermolysis: a new concept for cutaneous remodeling using microscopic patterns of thermal injury. Lasers Surg Med. 2004;34(5):426-38. doi: 10.1002/lsm.20048. PMID 15216537
- [Background] Brightman LA, Brauer JA, Anolik R, Weiss E, Karen J, Chapas A, Hale E, Bernstein L, Geronemus RG. Ablative and fractional ablative lasers. Dermatol Clin. 2009 Oct;27(4):479-89, vi-vii. doi: 10.1016/j.det.2009.08.009. PMID 19850197
- [Background] Hunzeker CM, Weiss ET, Geronemus RG. Fractionated CO2 laser resurfacing: our experience with more than 2000 treatments. Aesthet Surg J. 2009 Jul-Aug;29(4):317-22. doi: 10.1016/j.asj.2009.05.004. PMID 19717066
- [Background] Olsson MJ, Juhlin L. Long-term follow-up of leucoderma patients treated with transplants of autologous cultured melanocytes, ultrathin epidermal sheets and basal cell layer suspension. Br J Dermatol. 2002 Nov;147(5):893-904. doi: 10.1046/j.1365-2133.2002.04837.x. PMID 12410698
- [Background] Drake LA, Dinehart SM, Farmer ER, Goltz RW, Graham GF, Hordinsky MK, Lewis CW, Pariser DM, Skouge JW, Turner ML, Webster SB, Whitaker DC, Lowery BJ, Nordlund JJ, Grimes PE, Halder RM, Minus HR. Guidelines of care for vitiligo. American Academy of Dermatology. J Am Acad Dermatol. 1996 Oct;35(4):620-6. doi: 10.1016/s0190-9622(96)90691-x. No abstract available. PMID 8859294
- [Background] Njoo MD, Westerhof W. Vitiligo. Pathogenesis and treatment. Am J Clin Dermatol. 2001;2(3):167-81. doi: 10.2165/00128071-200102030-00006. PMID 11705094
- [Background] Taieb A, Picardo M. Clinical practice. Vitiligo. N Engl J Med. 2009 Jan 8;360(2):160-9. doi: 10.1056/NEJMcp0804388. No abstract available. PMID 19129529
- [Background] Hann SK, Lee HJ. Segmental vitiligo: clinical findings in 208 patients. J Am Acad Dermatol. 1996 Nov;35(5 Pt 1):671-4. doi: 10.1016/s0190-9622(96)90718-5. PMID 8912558
- [Background] Murakami T, Fukai K, Oiso N, Hosomi N, Kato A, Garganta C, Barnicoat A, Poppelaars F, Aquaron R, Paller AS, Ishii M. New KIT mutations in patients with piebaldism. J Dermatol Sci. 2004 Jun;35(1):29-33. doi: 10.1016/j.jdermsci.2004.03.003. PMID 15194144
- [Background] van Geel N, Wallaeys E, Goh BK, De Mil M, Lambert J. Long-term results of noncultured epidermal cellular grafting in vitiligo, halo naevi, piebaldism and naevus depigmentosus. Br J Dermatol. 2010 Dec;163(6):1186-93. doi: 10.1111/j.1365-2133.2010.10014.x. PMID 20804490
- [Background] Linthorst Homan MW, Spuls PI, de Korte J, Bos JD, Sprangers MA, van der Veen JP. The burden of vitiligo: patient characteristics associated with quality of life. J Am Acad Dermatol. 2009 Sep;61(3):411-20. doi: 10.1016/j.jaad.2009.03.022. Epub 2009 Jul 3. PMID 19577331
- [Background] Ongenae K, Van Geel N, De Schepper S, Naeyaert JM. Effect of vitiligo on self-reported health-related quality of life. Br J Dermatol. 2005 Jun;152(6):1165-72. doi: 10.1111/j.1365-2133.2005.06456.x. PMID 15948977
- [Background] Alikhan A, Felsten LM, Daly M, Petronic-Rosic V. Vitiligo: a comprehensive overview Part I. Introduction, epidemiology, quality of life, diagnosis, differential diagnosis, associations, histopathology, etiology, and work-up. J Am Acad Dermatol. 2011 Sep;65(3):473-491. doi: 10.1016/j.jaad.2010.11.061. PMID 21839315
- [Background] Fongers A, Wolkerstorfer A, Nieuweboer-Krobotova L, Krawczyk P, Toth GG, van der Veen JP. Long-term results of 2-mm punch grafting in patients with vitiligo vulgaris and segmental vitiligo: effect of disease activity. Br J Dermatol. 2009 Nov;161(5):1105-11. doi: 10.1111/j.1365-2133.2009.09367.x. Epub 2009 Jun 22. PMID 19673878
- [Background] Falabella R. Grafting and transplantation of melanocytes for repigmenting vitiligo and other types of leukoderma. Int J Dermatol. 1989 Jul-Aug;28(6):363-9. doi: 10.1111/j.1365-4362.1989.tb02479.x. No abstract available. PMID 2670786
- [Background] Gawkrodger DJ, Ormerod AD, Shaw L, Mauri-Sole I, Whitton ME, Watts MJ, Anstey AV, Ingham J, Young K; Therapy Guidelines and Audit Subcommittee, British Association of Dermatologists; Clinical Standards Department, Royal College of Physicians of London; Cochrane Skin Group; Vitiligo Society. Guideline for the diagnosis and management of vitiligo. Br J Dermatol. 2008 Nov;159(5):1051-76. doi: 10.1111/j.1365-2133.2008.08881.x. PMID 19036036
- [Background] Gawkrodger DJ, Ormerod AD, Shaw L, Mauri-Sole I, Whitton ME, Watts MJ, Anstey AV, Ingham J, Young K. Vitiligo: concise evidence based guidelines on diagnosis and management. Postgrad Med J. 2010 Aug;86(1018):466-71. doi: 10.1136/pgmj.2009.093278. PMID 20709768
- [Background] Malakar S, Dhar S. Treatment of stable and recalcitrant vitiligo by autologous miniature punch grafting: a prospective study of 1,000 patients. Dermatology. 1999;198(2):133-9. doi: 10.1159/000018089. PMID 10325459
- [Background] Boersma BR, Westerhof W, Bos JD. Repigmentation in vitiligo vulgaris by autologous minigrafting: results in nineteen patients. J Am Acad Dermatol. 1995 Dec;33(6):990-5. doi: 10.1016/0190-9622(95)90292-9. PMID 7490371
- [Background] Mulekar SV. Long-term follow-up study of segmental and focal vitiligo treated by autologous, noncultured melanocyte-keratinocyte cell transplantation. Arch Dermatol. 2004 Oct;140(10):1211-5. doi: 10.1001/archderm.140.10.1211. PMID 15492183
- [Background] Gravante G, Di Fede MC, Araco A, Grimaldi M, De Angelis B, Arpino A, Cervelli V, Montone A. A randomized trial comparing ReCell system of epidermal cells delivery versus classic skin grafts for the treatment of deep partial thickness burns. Burns. 2007 Dec;33(8):966-72. doi: 10.1016/j.burns.2007.04.011. Epub 2007 Sep 29. PMID 17904748
- [Background] Navarro FA, Stoner ML, Lee HB, Park CS, Wood FM, Orgill DP. Melanocyte repopulation in full-thickness wounds using a cell spray apparatus. J Burn Care Rehabil. 2001 Jan-Feb;22(1):41-6. doi: 10.1097/00004630-200101000-00009. PMID 11227683
- [Background] Wood FM, Giles N, Stevenson A, Rea S, Fear M. Characterisation of the cell suspension harvested from the dermal epidermal junction using a ReCell(R) kit. Burns. 2012 Feb;38(1):44-51. doi: 10.1016/j.burns.2011.03.001. Epub 2011 Nov 12. PMID 22079538
- [Background] Cervelli V, De Angelis B, Balzani A, Colicchia G, Spallone D, Grimaldi M. Treatment of stable vitiligo by ReCell system. Acta Dermatovenerol Croat. 2009;17(4):273-8. PMID 20021980
- [Background] Cervelli V, Spallone D, Lucarini L, Palla L, Brinci L, De Angelis B. Treatment of stable vitiligo hands by ReCell system: a preliminary report. Eur Rev Med Pharmacol Sci. 2010 Aug;14(8):691-4. PMID 20707289
- [Background] Chernoff G, Slatkine M, Zair E, Mead D. SilkTouch: a new technology for skin resurfacing in aesthetic surgery. J Clin Laser Med Surg. 1995 Apr;13(2):97-100. doi: 10.1089/clm.1995.13.97. PMID 10150575
- [Background] Hantash BM, Bedi VP, Chan KF, Zachary CB. Ex vivo histological characterization of a novel ablative fractional resurfacing device. Lasers Surg Med. 2007 Feb;39(2):87-95. doi: 10.1002/lsm.20405. PMID 17115384
- [Background] Gauthier Y, Surleve-Bazeille JE. Autologous grafting with noncultured melanocytes: a simplified method for treatment of depigmented lesions. J Am Acad Dermatol. 1992 Feb;26(2 Pt 1):191-4. doi: 10.1016/0190-9622(92)70024-a. PMID 1552051
- [Background] Ragland HP, McBurney E. Complications of resurfacing. Semin Cutan Med Surg. 1996 Sep;15(3):200-7. doi: 10.1016/s1085-5629(96)80051-4. PMID 8948539
- [Background] Wind BS, Meesters AA, Kroon MW, Beek JF, van der Veen JP, Nieuweboer-Krobotova L, Bos JD, Wolkerstorfer A. Punchgraft testing in vitiligo; effects of UVA, NB-UVB and 632.8 nm Helium-Neon laser on the outcome. J Eur Acad Dermatol Venereol. 2011 Oct;25(10):1236-7. doi: 10.1111/j.1468-3083.2010.03874.x. Epub 2010 Oct 6. No abstract available. PMID 21039919
- [Background] Linthorst Homan MW, Wolkerstorfer A, Sprangers MA, van der Veen JP. Digital image analysis vs. clinical assessment to evaluate repigmentation after punch grafting in vitiligo. J Eur Acad Dermatol Venereol. 2013 Feb;27(2):e235-8. doi: 10.1111/j.1468-3083.2012.04568.x. Epub 2012 May 23. PMID 22621363